CLINICAL TRIAL: NCT04003883
Title: ST-T Segment Changes in Emergency Physicians While on Duty
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Mathias Maleczek, Registrar, Medical University of Vienna
Other Study IDs: 1646/2019
Record Dates: First submitted 2019-06-25; First posted 2019-07-01 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: ST-T Segment Changes
Keywords: ST segment; preclinical emergency medicine; stress; occupational health; emergency medicine; 24h ECG
MeSH Terms: interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Emergency physicians: Emergency physicians doing shifts at the Medical University of Vienna's emergency response car will recieve a thorough cardiac pretesting. During shifts they will be attached to a Holter-ECG to detect changes in ST-T Segment and other ECG changes. Furthermore surrogate parameters of stress will be measured
  Interventions: Device: Holter ECG

INTERVENTIONS:
Device: Holter ECG — A Holter ECG will be recorderd during shifts

SUMMARY:
Preclinical emergency management is frequently associated with a combination of physical and psychological stress.

This stress is known to lead to a broad variety of changes in the physiology even extending in the cardiovascular system. Both physical and psychological stress induces ECG changes. These changes include not only arrhythmias but also deviations in ST-T segment representing the phase of repolarization.

Information about changes in ST-T segment are missing until now. The investigators hypothesise that ST-T deviations occur in emergency physicians during shift at an emergency response car.

In order to show changes in ST-T segment a prospective observational trial will be conducted. By using a 12 lead ECG Holter the investigators will obtain ECGs during shifts of emergency physicians at an emergency response vehicle.

During 12-hour shifts emergency physicians will be attached to the 12 lead Holter ECG. ECGs will be analysed after blinding of names and reason of call (code) to the investigators. The primary outcome will be ST-T segment changes greater than 0.1mV in two corresponding leads for more than 30 seconds per 100 calls.

As secondary outcomes, other ECG changes such as ST-T segment changes <0.1mV, T wave inversion or HRV will be analysed. Furthermore, surrogate parameter of stress will be measured using NASA-Task Load Index and cognitive appraisal and correlated to ST-T segment changes. Correlations between different phases of calls, different indications of calls and ECG changes will be assessed. Furthermore, correlation between alarm codes apriori defined as stressfull using a delphi process and ST-T segment changes as well es surrogate parameters of stress will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy emergency physicians doing shifts at the Medical University of Vienna's emergency response car

Exclusion Criteria:

* Known pregnancy
* Pre-existing cardiac diseases (valvular heart disease > I°, any form of cardiomyopathy, history of coronary artery disease, history of myocarditis, any channelopathy, known high degree (>1% of all beats within 24h) premature atrial or ventricular beats or atrial fibrillation or conduction disturbance.
* Any antiarrhythmic therapy
* Any implanted cardiac device
* Manifest Hyperthyroidism
* Termination of exercise testing due to the commonly used criteria26 or not reaching 85% of maximal predicted load.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Emergency physicians working at the Medical University of Vienna's emergency response cars will be invited to take part in this trial. Participants will be recruited by personalised phone contact, via email or direct approach and will not financially benefit for participation. The emergency physicians are anaesthesiologists and emergency medicine consultants and senior anaesthesia or emergency medical residents with prehospital emergency medicine credentials.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
ST-T segment change | Day1-3
  ST-T segment changes of at least 0.1mV in two corresponding leads occurring for more than 30 seconds per 100 prehospital emergency response calls

SECONDARY OUTCOMES:
ST-T segment change <0.1mV, <30sec. | Day1-3
T wave inversion > 30sec. | Day1-3
T wave inversion <= 30sec. | Day1-3
Changes in HRV | Day1-3
  Changes in HRV (SDNN, r-MSSD and pNN50) during calls compared to a baseline of 10min rest recorded at the beginning of shift as an emergency physician
Association of different phases of a call to changes in ST-T segments > 0.1mV in two corresponding leads for > 30sec. | Day1-3
Association of different phases of a call to changes in HRV (SDNN, r-MSSD and pNN50) | Day1-3
Association of the ten most stressful alarm codes to changes in ST-T segments > 0.1mV in two corresponding leads for > 30sec. | Day1-3
Association of the ten most stressful alarm codes to changes in HRV (SDNN, r-MSSD and pNN50) | Day1-3
Psychological stress during calls by means of NASA TLX | Day1-3
Frequency of calls being perceived as threat by using cognitive appraisal testing | Day1-3
Association of stressful and non-stressful calls to psychological stress measured using NASA TLX | Day1-3
Association of stressful and non-stressful calls to cognitive appraisal and calls that are perceived as threat. | Day1-3
Correlation of events logged | Day1-3
  Correlation of events logged by the emergency physician (treating a child, managing polytrauma, being woken up by the alarm, experiencing chest pain, performing an intubation or giving i.v. medication) to ST-T segment changes > 0.1mV in two corresponding leads for > 30sec.
Association of NASA TLX to ST-T segment changes > 0.1mV in two corresponding leads for > 30sec. | Day1-3
Association of cognitive appraisal to ST-T segment changes > 0.1mV in two corresponding leads for > 30sec. | Day1-3

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Maleczek, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maleczek M, Schebesta K, Hamp T, Burger AL, Pezawas T, Krammel M, Roessler B. ST-T segment changes in prehospital emergency physicians in the field: a prospective observational trial. Scand J Trauma Resusc Emerg Med. 2022 Jul 15;30(1):47. doi: 10.1186/s13049-022-01033-1. PMID 35841049